CLINICAL TRIAL: NCT04923789
Title: A Clinical Study to Evaluate the Efficacy and Safety of Autologous Hematopoietic Stem Cell Transplantation(ASCT) Bridging Chimeric Antigen Receptor T(CART) Cell Therapy in the Treatment of Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: A Study of ASCT Bridging CART Cell Therapy in Relapsed/Refractory B-cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020173
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2020-08

CONDITIONS: Relapsed Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASCT Without CART: Patients who undergone ASCT successfully and did not receive CART cell infusion.
- ASCT Bridging CART: Patients who undergone ASCT and received CART cell infusion sequently within 1 month. Patients with disease recurrence or progression prior to the infusion of CART cells will be excluded.

SUMMARY:
This is a single center, prospective cohort study to to evaluate the efficacy and safety of autologous hematopoietic stem cell transplantation(ASCT) bridging chimeric antigen receptor T (CART) cell therapy in the treatment of relapsed/refractory B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
High-dose chemotherapy followed by autologous hematopoietic stem cell transplantation(ASCT) is still the standard salvage treatment for relapsed/refractory B-cell non-Hodgkin's lymphoma (R/R B-NHL). However, its overall survival (OS) and event-free survival (EFS) of 3 years and above are less than 50%. Chimeric antigen receptor T (CART) cell therapy has shown great efficacy in treating B-NHL in recent years. Preclinical studies have indicated that the infusion of hematopoietic stem cells could promote the amplification and function of adoptive metastatic anti-tumor CD8+T cells, providing a certain theoretical basis for ASCT combined with CART cell therapy. In order to evaluate the efficacy and safety of ASCT bridging CART cell therapy in treating R/R B-NHL, we conduct this single center, prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed B-NHL with extrinsic involvement.
2. Age ≥ 18 years and ≤ 65 years.
3. Measurable disease of at least 15mm(node)/10mm（extranodal）
4. Meet any of the following conditions :1. After 4 courses of standard first-line treatment or 2 courses of treatment with more than two lines, the lesions decreased by less than 50%;2 B-NHL with disease progression after first-line or induction treatment;3. Relapsed B-NHL within 12 months after ASCT;4. After standard chemotherapy or hematopoietic stem cell transplantation, the size of any new lesions or the previously involved site which had achieved complete remission increased by 50% or more.
5. Receive standard autologous hematopoietic stem cell transplantation with CD34+ cells ≥2*10^6/kg.
6. Estimated survival time ≥3 months

Exclusion Criteria:

1. Having received allogeneic hematopoietic stem cell transplantation previously;
2. HIV-positive;
3. Active hepatitis B or C infection;
4. Previous history of other malignant tumors. Excluded: Patients who had cured basal or squamous cell carcinoma of the skin and carcinoma in situ of the cervix at any time prior to the study; Patients with disease-free survival ≥5 years who had been cured by surgery only without further treatment for the other tumors listed above can be included in the study.
5. Patients with cardiac insufficiency:ejection fraction (EF) < 30%, NYHA standard, grade II or above
6. Patients with liver and renal insufficiency: Serum Direct Bilirubin (SB) ≥2mg/ dL (34.2μmol/L), Aspartate Aminotransferase(AST) > 2.5 times the up, Serum Creatinine (SCR) > 2.5mg/ dL (221μmol/L)
7. Female patients who are pregnant, preparing to become pregnant or lactating.
8. The investigator believes that there are other factors that are not suitable for inclusion or affect subjects' participation or completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The total number of patients was 60.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival(PFS) | up to 12 months
  The last follow-up of a surviving patient after ASCT to the date of relapse, disease progression, death, dependent upon which occurred first over a follow-up period of 18 months.
Overall Survival(OS) | up to 12 months
  The interval from the time of ASCT to death from any cause or to the last follow-up moment.

SECONDARY OUTCOMES:
Duration of Response(DOR) | up to 12 months
  DOR will be assessed from ASCT to progression,death or last follow-up.
Adverse Events(AE) | Measured from start of treatment until 28 days after last treatment.
  Number of participants with adverse events. Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 will be tabulated
Overall Response Rate(ORR) | up to 12 months
  Number of patients who achieved response after the treatment.
Cumulative Recurrence Rate | up to 12 months
  Cumulative number of patients who recurred after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China